CLINICAL TRIAL: NCT02124213
Title: Open Label Adaptive Design Study To Evaluate D1 Receptor Occupancy (ro) Following Single Dose Of Pf-06412562, Using Positron Emission Tomography (Pet) With Ligand [11c]sch23390 In Healthy Male Subjects
Brief Title: A Study To Evaluate D1 Receptor Occupancy (RO) Following Single Dose of PF-06412562 In Healthy Male Volunteers
Acronym: PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7441005; 2013-004356-37 (EudraCT Number)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Receptor Occupancy; PET; D1 Receptor Agonist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohor 1 - 30 mg (Experimental): Cohort will include approximately 4 HVs/completers who will receive a single 30 mg dose of PF-06412562.
  Interventions: Drug: 30 mg PF-06412562
- Cohort 2 ( adaptive dose, optional) (Experimental): Cohort 2 will include approximately 4 HVs/completers who will receive a single dose of PF-06412562. The dose will be selected based on the results obtained for Cohort 1.
  Interventions: Drug: PF-06412562
- Cohort 3 ( adaptive dose, optional) (Experimental): Cohort 2 will include approximately 4 HVs/completers who will receive a single dose of PF-06412562. The dose will be selected based on the results obtained for Cohort 1 and Cohort 2.
  Interventions: Drug: PF-06412562

INTERVENTIONS:
Drug: 30 mg PF-06412562 — Subject will receive a single dose of 30 mg PF-06412562
  Arms: Cohor 1 - 30 mg
Drug: PF-06412562 — The dose will be selected based on the results obtained for Cohort 1. This Cohort is optional.
  Arms: Cohort 2 ( adaptive dose, optional)
Drug: PF-06412562 — The dose will be selected based on the results obtained for Cohort 1 and Cohort 2.
  This Cohort is optional.
  Arms: Cohort 3 ( adaptive dose, optional)

SUMMARY:
This study will evaluate D1 Receptor Occupancy (RO) following a single dose of PF-06412562 In healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

Healthy Male Volunteers

Exclusion Criteria:

Evidence or history of clinically significant hepatic, renal, cardiovascular, endocrine, hematologic, gastrointestinal, pulmonary, neurologic, oncologic, psychiatric, or allergic disease Any condition possibly affecting drug absorption A positive urine drug screen

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
PF-06142562 plasma exposure and RO in the striatum | Day 1
  Using Positron Emission Tomography and a radiotracer [11C]SCH23390, the PF-06142562 plasma exposure and RO in the striatum (average of caudate and putamen) will be measured in healthy male subjects.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 1
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Day 1
Area under the plasma concentration-time profile from time zero to the last plasma measurement at 4 hours (AUC0-4) | Day 1
Average plasma concentration over 4 hours (Cav,0-4) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Karolinska Trial Alliance (KTA) M62, Huddinge, Stockholm County, Sweden

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7441005&StudyName=A%20Study%20To%20Evaluate%20D1%20Receptor%20Occupancy%20%28RO%29%20Following%20Single%20Dose%20of%20PF-06412562%20In%20Healthy%20Male%20Volunteers